CLINICAL TRIAL: NCT07126236
Title: Response-adaptive to Epcoritamab In First Relapse: A Phase II, Response-adaptive, Open-Label, Multicenter Study to Evaluate the Efficacy of Eptoritamab in Patients With Relapse/Refractory Large B Cell Lymphoma
Brief Title: Response-adaptive to Epcoritamab In First Relapse: Study to Evaluate the Efficacy of Eptoritamab in Patients With Relapse/Refractory Large B Cell Lymphoma
Acronym: REPIFIR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Collaborators: AbbVie (Industry); Incyte Corporation (Industry); Evidenze Health España (CRO) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REPIFIR-AGR-GEL-23; 2024-514440-86-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-10; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Large B Cell Lymphoma
Keywords: lymphoma; geltamo; DIFFUSE LARGE B-CELL LYMPHOMA; DLBCL; RELAPSE; epcoritamab; tafasitamab; lenalidomide
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Recurrence | interventions — tafasitamab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EPCO monotherapy (Experimental): Epcoritamab in monotherapy will be administred until cycle 12.
  Interventions: Drug: Epcoritamab
- Combination therapy (Experimental): 3 cycles of Epcoritamab in monotherapy will be administred and then Epcoritamab will be administred with Tafasitamab and Lenalidomide from cycle 4 until cycle 15.
  Interventions: Drug: Epcoritamab, tafasitamab and lenalidomide

INTERVENTIONS:
Drug: Epcoritamab — Patients will receive 12 cycles of Epcoritamab monotherapy.
  Arms: EPCO monotherapy
Drug: Epcoritamab, tafasitamab and lenalidomide — Patients will receive 3 cycles of Epcoritamab monotherapy and then 12 cycles of Epcoritamab, Tafasitamab and Lenalidomide.
  Arms: Combination therapy

SUMMARY:
phase II, response-adaptive, open-label, multicenter study aiming to include 80 patients in 78 months. Patients will receive 3 cycles of epcoritamab monotherapy and, since cycle 4, they can continue with epcoritamab monotherapy until cycle 12 or change to combination therapy (epcoritamab + tafasitamab + lenalidomide) until cycle 15. Patients will be followed up to 5 years.

DETAILED DESCRIPTION:
Epcoritamab is a full-length bispecific IgG1 antibody directed against two proteins, CD3 on the T lymphocyte and CD20 on the lymphoma cell. This antibody redirects and activates T cells, generating an immune synapse that eventually eliminates malignant cells expressing CD20.

Previous studies have demonstrated that Epcoritamab has potent antitumor activity as a monotherapy agent, with a favorable and manageable safety profile.

Since its efficacy is so favorable it is reasonable to think that it could be an excellent option for first-relapse patients. However, to date, there is no data on this therapy's usefulness as second-line treatment. Therefore we intend to evaluate the efficacy of Epcoritamab as a treatment option for patients with first-relapse LBCL.

The purpose of this study is to determine the efficacy of Epcoritamab as second line treatment for LBCL patients. On the basis of the clinical experience, it is hypothesized that Epcoritamab would provide a better complete response rate (CRR) in comparison to Platinum-based immunochemotherapy (CRR=25%), Polatuzumab-Bendamustin Rituximab (CRR=40%) and Tafasitamab-Lenalidomide (CRR=43%).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any study-specific assessment is performed.
2. Age >18 years
3. Patients with Relapse/Refractory histologically confirmed LBCL, including, Diffuse Large B Cell Lymphoma (DLBCL); Primary Mediastinal Large B Cell Lymphoma (PMBCL), High-grade B-cell lymphoma (HGBCL); and grade 3B Follicular Lymphoma.

   Relapsed disease is defined as complete remission to first line therapy followed by a recurrence of the disease after a minimum of 6 months of completion of first-line therapy. A biopsy at the time of relapse is recommended but not mandatory.

   Refractory disease is defined as no objective response to first line therapy (biopsy not mandatory if diagnostic sample available). Four groups of patients are eligible:
   * PD as best response to first line therapy.
   * SD as best response after at least 4 cycles of first line therapy.
   * PR as best response after at least 6 cycles of first line therapy.
   * CR and disease recurrence within < 6 months from the completion of first-line therapy.
4. Patients must have received adequate first-line therapy including at a minimum: an anti-CD20 monoclonal antibody (rituximab or obinutuzumab), and CHOP (cyclophosphamide, hydroxydaunomycin, oncovin, and prednisone) or CHOP-like chemotherapy.
5. At the investigator's discretion, the patient should not be a candidate for 1st relapse CAR-T therapy or unwilling to receive CAR-T therapy.
6. Patients must be autologous stem cell transplantation (ASCT)-ineligible: Age ≥65 and/or HTC-CI ≥3 or or unwilling to receive transplant.
7. PET positive disease.
8. Performance status according to Eastern Cooperative Oncology Group (ECOG) 0 to 2.
9. Patients meeting with the following hematology values:

   * Hemoglobin ≥8 g/dl (transfusion support permitted but not within 7 days of screening lab collection)
   * Absolute neutrophil count (ANC) ≥ 1/109/L (growth factor support allowed in case of bone marrow involvement).
   * Absolute lymphocyte count ≥ 0.1/109/L,
   * Platelet count ≥ 70/109/L (unless secondary to bone marrow involvement, OR ≥50x/109/L if documented bone marrow involvement). Platelet transfusions permitted but not within 7 days of screening lab collection.
10. Female patients of child-bearing potential must have a negative urine or serum pregnancy test at screening and agree to use highly effective methods of contraception (e.g., established use of oral, injected or implanted combined (estradiol and progesterone containing) hormonal contraception; placement of an intrauterine device (IUD) or intrauterine system (IUS) upon enrollment according to the recommendations provided by Clinical Trial Facilitation Group (CTFG), during the treatment period and for 4 months after the last dose of study medication. Moreover, the patient must agree to ongoing pregnancy testing during the course of the study, and after study therapy has ended. This applies even if the patient practices complete and continued sexual abstinence.

    Women not of childbearing potential are defined as: premenarchal; postmenopausal (greater than 50 years of age with amenorrhea for at least 12 months or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone (FSH) level greater than 40 IU per L or milli-International unit (mIU) per mL); permanently sterilized (e.g., bilateral tubal occlusion [which includes tubal ligation procedures as consistent with local regulations], hysterectomy, bilateral salpingectomy, bilateral oophorectomy); or otherwise be incapable of pregnancy.
11. Male patients must use a reliable method of contraception (if sexually active with a female of child-bearing potential) upon enrollment according to the recommendations provided by CTFG, during the treatment period, and for 4 months following the last dose of investigational drug or agreement to remain abstinent. Agreement to refrain from donating blood or sperm during the study participation and for 4 months after the last dose of study medication.
12. Women must agree not to donate blood or oocytes during the course of the study and for 4 months after the last dose of study medication. Restrictions concerning blood donation apply as well to females who are not of childbearing potential. Men must also not donate sperm during the trial and for 4 months after receiving the last dose of study drug.
13. Females of childbearing potential must refrain from breastfeeding during the course of the study and for 4 months after the last dose of study medication.
14. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
15. Not included in other clinical trial or treated with an experimental drug.

Exclusion Criteria:

1. Patients who received more than one prior line of systemic therapy
2. Patients with detectable Central Nervous System (CNS) lymphoma
3. Significant organ function impairment:

   * creatinine clearance calculated by Cockcroft-Gault ≤ 45 ml/min
   * direct bilirubin level < 2 x ULN (except in patients with Gilbert's syndrome),
   * alanine transaminase (ALT) and aspartate aminotransferase (AST) >3 × ULN or >5 × ULN in cases of documented liver involvement.
   * clinically relevant pleural effusion,
   * left ventricular ejection fraction (LVEF) ≤ 45%
4. Serious accompanying disorder leading to impaired organ function causing significant clinical problems and reduced life expectancy of less than 3 months.
5. Have a history of deep venous thrombosis/embolism, threatening thromboembolism or known thrombophilia or are at a high risk for a thromboembolic event in the opinion of the investigator and who are not willing/able to take venous thromboembolic event prophylaxis during the entire treatment period
6. Known clinically significant cardiac disease, including:

   * Onset of unstable angina pectoris within 6 months of signing the patient informed consent form.
   * Acute myocardial infarction within 6 months of signing the patient informed consent form.
   * Congestive heart failure (grade III or IV as classified by the New York Heart Association.
   * Left ventricular ejection fraction ≤45%.
7. Known past or current malignancy other than inclusion diagnosis, except for: Cervical carcinoma of Stage 1B or less; Non-invasive basal cell or squamous cell skin carcinoma; Non-invasive, superficial bladder cancer; Localized low grade prostate cancer (up to Gleason score 6); DCIS of the breast; Other malignancy that has been treated with curative intent and has remained in remission for 3 years.
8. Previous ASCT.
9. Prior anti-CD3 and CD20 bispecific antibodies therapy or prior treatment with tafasitamab.
10. Presence of severe infection that is uncontrolled or requiring IV antimicrobials for management.
11. History of HIV infection or acute or chronic active hepatitis B or C infection.

    * Individuals with positive HIV serology may be included if negative viral load and CD4 >200/mm3. For being included, patients should have controlled disease and been on treatment for at least 1 year
    * Individuals with history of hepatitis infection with positive antibodies (anti-HB and anti-HV) might be included if negative viral load (negative hepatitis B PCR). Patients who are HBcAb positive must receive HBV prophylaxis while on treatment. Patients with positive HbsAg are excluded. Patients who are hepatitis B PCR positive will be excluded. Patients who are hepatitis C RNA positive will be excluded.
12. Females who are pregnant or breastfeeding.
13. Richter's transformation or prior chronic lymphocytic leukemia (CLL).
14. Treatment with radiotherapy, chemotherapy, immunotherapy, immunosuppressive therapy, or any investigational agent for the purposes of treating cancer within 4 weeks prior to Cycle 1 Day 1.
15. Recent major surgery (within 4 weeks before the start of Cycle 1 Day 1) other than for diagnosis.
16. Vaccination with a live vaccine or COVID-19 vaccination within 4 weeks prior to treatment.
17. History of hypersensitivity to any of the study drugs or their ingredients or to drugs with similar structure. History of severe allergic or anaphylactic reactions to human, humanized, chimeric, or murine monoclonal antibodies.
18. Close affiliation with the investigator (e.g. a close relative) or persons working at the study site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Epcoritamab monotherapy | Cycle 3, cycle 4, cycle 7, cycle 10, cycle 13 (for combination therapy) and EoT (28 days after last administration of investigational product) visits. Each cycle is 28 days.
  The efficacy of Epcoritamab monotherapy will be centrally evaluated by the best CRR at any moment since initiation. The CRR will be assessed by PET-CT according to Lugano Classification and is defined as the proportion of patients who achieve a best response of complete response (CR) at any moment since initiation of Epcoritamab first administration.

SECONDARY OUTCOMES:
Efficacy of Epcoritamab monotherapy after 3 cycles | At the end of cycle 3 (each cycle is 28 days)
  The efficacy of Epcoritamab monotherapy will be centrally evaluated by the best CRR, defined as the proportion of patients who achieve a best response of CR after 3 cycles of Epcoritamab administration.
Efficacy of Epcoritamab monotherapy and combination therapy by CRR | Cycle 3, cycle 4, cycle 7, cycle 10, cycle 13 (for combination therapy) and EoT (28 days after last administration of investigational product) visits. Each cycle is 28 days.
  The efficacy of Epcoritamab monotherapy and combination therapy with tafasitamab-lenalidomide will be evaluated by local investigators and central evaluation as per CRR (locally evaluated for Epcoritamab monotherapy; local and central evaluation for combination therapy).
Evaluation of MRD | Cycles 3, 4, 7, 10, 12, 13, 15 (each cycle is 28 days), EoT (28 days after last administration of Study drug) and cycles 18 and 24 (epcoritamab monotherapy) or cycles 21 and 27 (combination therapy) visits (each cycle is 28 days).
  The efficacy of Epcoritamab monotherapy and combination therapy will be evaluated by MRD (positive or negative) from ctDNA samples immediately before initiation of C3, C4, C7, C10, C12, C13, C15, End of Treatment (EoT) and cycles 18/24 (epcoritamab monotherapy) or cycles 21/27 (combination therapy).
Evaluation of patients with negative MRD by PFS | At cycle 3 visit (each cycle is 28 days).
  The PFS of patients with negative MRD at Visit 3 (V3) (immediately before administrating C3 of Epcoritamab monotherapy).
Safety and tolerability | Baseline, during all the cycles day 1 visit (each cycle is 28 days) and at EoT (28 days afert las administration of Study drug).
  The safety and tolerability of Epcoritamab monotherapy and combination therapy are evaluated as follows:
  * Type, frequency, and severity of adverse events (AEs).
  * Type, frequency, and severity of Adverse events of special interest (AESIs): Cytokine release syndrome (CRS), immune effector cell-associated neurotoxicity syndrome (ICANS), clinical tumor lysis syndrome (CTLS) and other safety topics of interest (tumour flare reaction, prolonged cytopenia, serious infections and second primary malignancies).
  * Incidence, severity, and treatment.
Efficacy of Epcoritamab Monotherapy and Combination therapy by ORR | Cycle 3, cycle 4, cycle 7, cycle 10, cycle 13 (for combination therapy) and EoT (28 days after last administration of investigational product) visits. Each cycle is 28 days
  The efficacy of Epcoritamab monotherapy and combination therapy with tafasitamab-lenalidomide will be evaluated by local investigators and central evaluation as per ORR at any time.
Efficacy of Epcoritamab Monotherapy and combination therapy by DoR | Cycle 3, cycle 4, cycle 7, cycle 10, cycle 13 (for combination therapy) and EoT (28 days after last administration of investigational product) visits. Each cycle is 28 days
  The efficacy of Epcoritamab monotherapy and combination therapy with tafasitamab-lenalidomide will be evaluated by local investigators and central evaluation as per DoR at any time.
Efficacy of Epcoritamab monotherapy and combination therapy by DoCR | Cycle 3, cycle 4, cycle 7, cycle 10, cycle 13 (for combination therapy) and EoT (28 days after last administration of investigational product) visits. Each cycle is 28 days
  The efficacy of Epcoritamab monotherapy and combination therapy with tafasitamab-lenalidomide will be evaluated by local investigators and central evaluation as per DoCR at any time.
Efficacy of Epcoritamab monotherapy and combination therapy by EFS | Cycle 3, cycle 4, cycle 7, cycle 10, cycle 13 (for combination therapy) and EoT (28 days after last administration of investigational product) visits. Each cycle is 28 days
  The efficacy of Epcoritamab monotherapy and combination therapy with tafasitamab-lenalidomide will be evaluated by local investigators and central evaluation as per Event-free survival (EFS) at any time.
Efficacy of Epcoritamab monotherapy and combination therapy by PFS | Cycle 3, cycle 4, cycle 7, cycle 10, cycle 13 (for combination therapy) and EoT (28 days after last administration of investigational product) visits. Each cycle is 28 days
  The efficacy of Epcoritamab monotherapy and combination therapy with tafasitamab-lenalidomide will be evaluated by local investigators and central evaluation as per PFS at any time.
Efficacy of Epcoritamab montherapy and combination therapy by OS | Cycle 3, cycle 4, cycle 7, cycle 10, cycle 13 (for combination therapy) and EoT (28 days after last administration of investigational product) visits. Each cycle is 28 days
  The efficacy of Epcoritamab monotherapy and combination therapy with tafasitamab-lenalidomide will be evaluated by local investigators and central evaluation as per OS at any time.
Evaluation of patients with negative MRD by OS | At cycle 3 visit (each cycle is 28 days).
  The OS of patients with negative MRD at Visit 3 (V3) (immediately before administrating C3 of Epcoritamab monotherapy).
Evaluation of patients with negative MRD by DoR | At cycle 3 visit (each cycle is 28 days).
  The DoR of patients with negative MRD at Visit 3 (V3) (immediately before administrating C3 of Epcoritamab monotherapy).

OTHER OUTCOMES:
Response of patients stopping treatment by PFS | At EoT visit (28 days after last administration of Study drug) for monotherapy and at C13 visit for combination therapy (each cycle is 28 days).
  To compare the PFS of patients stopping therapy after 1 year of treatment (CR by PET-CT and negative MRD) with the groups of patients who continue monotherapy or receive combination.
Correlation between biomarkers and study treatment by ORR | Cycles 3, 4, 7, 10, 12, 13, 15 (each cycle is 28 days), EoT (28 days after last administration of Study drug) and cycles 18 and 24 (epcoritamab monotherapy) or cycles 21 and 27 (combination therapy) visits (each cycle is 28 days).
  Correlation between biomarkers and study treatment efficacy determined by ORR.
Efficacy of Epcoritamab monotherapy and combination therapy in patients reintroducing treatment by DoR | After reintroduction of study treatment due to MRD positive result, on cycles 13, 16, 19, 22, 25, 28 visits (each cycle is 28 days).
  Efficacy of Epcoritamab or Epcoritamab/Tafasitamab by DoR in patients reintroducing the study treatment with a MRD positive result.
MRD negativity | through study completion, an average of 5 years
  Median duration of molecular response (MRD negativity).
Correlation between tumor volume and efficacy | Cycle 3, cycle 4, cycle 7, cycle 10, cycle 13 (for combination therapy) and EoT (28 days after last administration of investigational product) visits. Each cycle is 28 days.
  Correlation between Total Metabolic Tumor Volume (centrally evaluated) and study treatment efficacy determined by PFS and OS.
ctDNA levels | Cycles 3, 4, 7, 10, 12, 13, 15 (each cycle is 28 days), EoT (28 days after last administration of Study drug) and cycles 18 and 24 (epcoritamab monotherapy) or cycles 21 and 27 (combination therapy) visits (each cycle is 28 days).
  Descriptive analysis of dynamic changes in ctDNA levels
Correlation between lymphocyte subsets and efficacy | Through study completion, an average of 5 years.
  Correlation between lymphocyte subsets and study treatment efficacy determined by ORR, CRR, DoR, PFS and OS and safety determined by type, frequency, and severity of adverse events.
Response of patients stopping treatment | At EoT visit (28 days after last administration of Study drug) for monotherapy and at C13 visit for combination therapy (each cycle is 28 days).
  To compare the DoR of patients stopping therapy after 1 year of treatment (CR by PET-CT and negative MRD) with the groups of patients who continue monotherapy or receive combination.
Correlation between biomarkers and study treatment efficacy by CRR | Cycles 3, 4, 7, 10, 12, 13, 15 (each cycle is 28 days), EoT (28 days after last administration of Study drug) and cycles 18 and 24 (epcoritamab monotherapy) or cycles 21 and 27 (combination therapy) visits (each cycle is 28 days).
  Correlation between biomarkers and study treatment efficacy determined by CRR.
Correlation between biomarkers and study treatment efficacy DoR | Cycles 3, 4, 7, 10, 12, 13, 15 (each cycle is 28 days), EoT (28 days after last administration of Study drug) and cycles 18 and 24 (epcoritamab monotherapy) or cycles 21 and 27 (combination therapy) visits (each cycle is 28 days).
  Correlation between biomarkers and study treatment efficacy determined by DoR, PFS and OS.
Correlation between biomarkers and study treatment efficacy by PFS | Cycles 3, 4, 7, 10, 12, 13, 15 (each cycle is 28 days), EoT (28 days after last administration of Study drug) and cycles 18 and 24 (epcoritamab monotherapy) or cycles 21 and 27 (combination therapy) visits (each cycle is 28 days).
  Correlation between biomarkers and study treatment efficacy determined by PFS.
Correlation between biomarkers and study treatment efficacy by OS | Cycles 3, 4, 7, 10, 12, 13, 15 (each cycle is 28 days), EoT (28 days after last administration of Study drug) and cycles 18 and 24 (epcoritamab monotherapy) or cycles 21 and 27 (combination therapy) visits (each cycle is 28 days).
  Correlation between biomarkers and study treatment efficacy determined by OS.
Efficacy of Epcoritamab monotherapy and combination therapy in patients reintroducing treatment by PFS | After reintroduction of study treatment due to MRD positive result, on cycles 13, 16, 19, 22, 25, 28 visits (each cycle is 28 days)
  Efficacy of Epcoritamab or Epcoritamab/Tafasitamab by PFS in patients reintroducing the study treatment with a MRD positive result.
Efficacy of Epcoritamab monotherapy and combination therapy in patients reintroducing treatment by OS | After reintroduction of study treatment due to MRD positive result, on cycles 13, 16, 19, 22, 25, 28 visits (each cycle is 28 days)
  Efficacy of Epcoritamab or Epcoritamab/Tafasitamab by OS in patients reintroducing the study treatment with a MRD positive result.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Bastos-Oreiro, Principal Investigator — Hospital General Universitario Gregorio Marañón; Pau Abrisqueta, Principal Investigator — Hospital Universitari Vall d'Hebrón
Locations (15):
- Spain (15):
  - Hospital Universitario Miguel Servet, Zaragoza, Aragon
  - Hospital Universitario de Burgos, Burgos, Castille and León
  - ICO Badalona, Badalona, Catalonia
  - Hospital Universitari Vall d'Hebrón, Barcelona, Catalonia
  - Hospital San Pedro de Alcántara, Cáceres, Extremadura
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Universitario Infanta Leonor, Madrid, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitario Costa del Sol, Marbella, Málaga
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital Universitario Dr. Peset, Valencia, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia, Valencia
  - Hospital Universitario de Basurto, Bilbao, Vizcaya

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in hematology diseases. All individual data collected during the trial will be available. Data shared will be coded, with no PHI included. Study protocol, statistical analysis plan, informed consent form and clinical study report will be also available. Information will be available beginning 6 months after final publication with no end date established. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party. Data requests can be submitted starting 6 months after article publication. Access to trial IPD can be requested by qualified researchers and will be provided following review and approval of a research and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact to GELTAMO though the web page: https://www.geltamo.com/contacto

REFERENCES:
- See also: GELTAMO web page — https://www.geltamo.com/